CLINICAL TRIAL: NCT02745158
Title: FOP Connection: A Global Registry for the Fibrodysplasia Ossificans Progressiva Community
Brief Title: The Fibrodysplasia Ossificans Progressiva (FOP) Connection Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The International FOP Association (Other)
Responsible Party: Sponsor
Other Study IDs: IFOPA-REG-001
Record Dates: First submitted 2016-03-06; First posted 2016-04-20 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2016-03

CONDITIONS: Fibrodysplasia Ossificans Progressiva (FOP)
Keywords: Fibrodysplasia ossificans progressiva; FOP; International FOP Association; Patient Advocacy Group; Patient Registry; Natural History; Patient-Reported Outcomes; Observational Database; Bone Morphogenetic Protein; BMP; Bone Growth; Joint; Mobility; Flare-Up; Heterotopic Ossification; Ectopic Bone; Osteochondroma; Hallux Valgus; ALK2; ACVR1; Activin A; IFOPA; Activin A Receptor Type I; Activin Receptor-like Kinase-2
MeSH Terms: conditions — Myositis Ossificans; Ossification, Heterotopic; Osteochondroma; Hallux Valgus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FOP Patients

SUMMARY:
The Fibrodysplasia Ossificans Progressiva (FOP) Connection Registry is a global, non-interventional, voluntary database that captures demographic and disease data directly from FOP patients and their caregivers via a secure, web-based patient portal. A physician portal (in development) will allow physicians to enter clinical data about their patients. The objectives are to organize the international FOP community for participation in clinical trials; to enable FOP patients worldwide to report data in a shared forum; to improve the collective understanding of FOP natural history; and to advance the understanding of FOP treatment outcomes.

DETAILED DESCRIPTION:
The FOP Connection Registry is a global, non-interventional, voluntary database that captures demographic and disease data directly from FOP patients and their caregivers via a secure, web-based patient portal. No experimental intervention is involved. The objectives are to organize the international FOP community for participation in clinical trials; to enable FOP patients worldwide to report data in a shared forum; to improve the collective understanding of FOP natural history; and to advance the understanding of FOP treatment outcomes.

The Registry collects data through two sources. First, the Patient Portal (launched in July 2015) allows FOP patients and caregivers to enter information about their experiences living with FOP. Second, the Physician Portal (in development) will allow physicians to enter clinical data about patients under their care. The Registry will be capable of including data on specific marketed therapies under the direction and control of a sponsoring pharmaceutical company. Key identifiers will link the physician-reported data with the Patient Portal data.

Participants must have a confirmed diagnosis of FOP and the participant (or a parent or legal guardian) must be willing and able to provide written informed consent. There are no exclusion criteria. Data collected in the Patient Portal include: patient demographics and diagnosis pathway; medical and dental care; clinical research participation and biospecimen donation; heterotopic ossification (bone growth and episodic flare-ups); other signs and symptoms by body system; patient-reported outcomes (physical functioning, pain, fatigue, and general health); and assistive devices, aids, attendants, and adaptations. Because the Registry is designed to accommodate participants along a broad spectrum of FOP disease severity, most of the data fields are optional, allowing participants a high degree of flexibility in how much information they contribute, which also minimizes participant burden.

After completing the informed consent, participants enter their baseline (historical) data. Participants will be encouraged to update their information at least twice per year. Participants may withdraw their consent at any time without prejudice or providing an explanation. The Registry has no pre-specified end date and will continue for as long as it is sustainable and useful to the FOP community.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a confirmed diagnosis of FOP.
* Participants (or a parent or legal guardian) must be willing and able to provide written informed consent.

Exclusion Criteria:

* There are no exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with Fibrodysplasia Ossificans Progressive (FOP) from the international FOP community will be invited to join the Registry.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Changes in New Bone Growth Using a Patient-Directed Survey Developed by the IFOPA | Baseline, then every six months for up to 10 years
  The patient is able to report changes in new bone growth among 27 joints and body locations.
Patient Reported Changes in Episodic Flare-Ups Using a Patient-Directed Survey Developed by the IFOPA | Baseline, then every six months for up to 10 years
  The patient is able to report changes in episodic flare-ups among 27 joints and body locations.
Patient Reported Changes in Mobility Using a Patient-Directed Survey Developed by the IFOPA | Baseline, then every six months for up to 10 years
  The patient is able to report changes in mobility among 27 joints and body locations.

SECONDARY OUTCOMES:
Patient Reported Changes in Health Resource Utilization Using a Patient-Directed Survey Developed by the IFOPA | Baseline, then every six months for up to 10 years
  The number of visits to a Physician and a Dentist, as well as the number of hospitalizations and reasons for the hospitalizations, are used to assess health resource utilization.
Patient Reported Changes in Signs Related to the Ear Using a Patient-Directed Survey Developed by the IFOPA | Baseline, then every six months for up to 10 years
  The patient is able to report new or continuing health issues related to the ears.
Patient Reported Changes in Signs Related to the Skin Using a Patient-Directed Survey Developed by the IFOPA | Baseline, then every six months for up to 10 years
  The patient is able to report new or continuing health issues related to the skin.
Patient Reported Changes in Signs Related to the Central Nervous System Using a Patient-Directed Survey Developed by the IFOPA | Baseline, then every six months for up to 10 years
  The patient is able to report new or continuing health issues related to the central nervous system.
Patient Reported Changes in Signs Related to the Pulmonary System Using a Patient-Directed Survey Developed by the IFOPA | Baseline, then every six months for up to 10 years
  The patient is able to report new or continuing health issues related to the pulmonary system.
Patient Reported Changes in Signs Related to the Gastrointestinal System Using a Patient-Directed Survey Developed by the IFOPA | Baseline, then every six months for up to 10 years
  The patient is able to report new or continuing health issues related to the gastrointestinal system.
Patient Reported Changes in Signs Related to the Cardiovascular System Using a Patient-Directed Survey Developed by the IFOPA | Baseline, then every six months for up to 10 years
  The patient is able to report new or continuing health issues related to the cardiovascular system.
Patient Reported Changes in Signs Related to the Renal System Using a Patient-Directed Survey Developed by the IFOPA | Baseline, then every six months for up to 10 years
  The patient is able to report new or continuing health issues related to the renal system.
Patient Reported Changes in Signs Related to the Endocrine System Using a Patient-Directed Survey Developed by the IFOPA | Baseline, then every six months for up to 10 years
  The patient is able to report new or continuing health issues related to the endocrine system.

OTHER OUTCOMES:
Patient Reported Changes in Activities of Daily Living Using the FOP-Physical Functioning Questionnaire (PFQ) | Baseline, then every six months for up to 10 years
Patient Reported Changes in Overall Health Using the PROMIS Global Health Scale | Baseline, then every six months for up to 10 years
Patient Reported Changes in the Need for Assistive Devices, Aids, Attendants, and Adaptations Using a Survey Developed by the IFOPA | Baseline, then every six months for up to 10 years
  The patient is able to respond Yes or No to questions related to his/her need for Assistive Devices, Aids, Attendants, and Adaptations as a result of his/her FOP disease.

CONTACTS AND LOCATIONS:
Overall Officials: Betsy Bogard, BS, MS, Study Director — The International FOP Association
Locations (1):
- The International FOP Association, Casselberry, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Formal data sharing agreements are planned between the International FOP Association and biopharmaceutical companies doing research in Fibrodysplasia Ossificans Progressiva (FOP). Publications are also planned with biopharmaceutical companies and physician researchers.

REFERENCES:
- [Derived] Pignolo RJ, Kimel M, Whalen J, Kawata AK, Artyomenko A, Kaplan FS. The Fibrodysplasia Ossificans Progressiva Physical Function Questionnaire (FOP-PFQ): A patient-reported, disease-specific measure. Bone. 2023 Mar;168:116642. doi: 10.1016/j.bone.2022.116642. Epub 2022 Dec 13. PMID 36526263
- See also: Click here for more information about this study: The FOP Connection Registry — http://www.fopconnection.org
- See also: The International FOP Association is a 501(c)(3) non-profit organization supporting medical research, education and communication for those afflicted by the rare genetic condition Fibrodysplasia Ossificans Progressiva (FOP). — http://www.ifopa.org